CLINICAL TRIAL: NCT04166669
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study of APX001 to Evaluate the Effects of CYP3A4 Inhibition and Pan-CYP Induction in Two Parallel Groups of Healthy Male and Female Subjects
Brief Title: A Drug-Drug Interaction Study of CYP3A4 Inhibition and Pan-CYP Induction on APX001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APX001-107; C4791007 (Other: Alias Study Number)
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Drugs: APX001, itraconazole
  Interventions: Drug: APX001; Drug: Itraconazole
- Cohort 2 (Experimental): Drugs: APX001, rifampin
  Interventions: Drug: APX001; Drug: Rifampin

INTERVENTIONS:
Drug: APX001 — Cohort 1 Day 1: APX001 500 mg IV BID over a 3-hour infusion; Day 18: APX001 500 mg IV BID over a 3-hour infusion. Cohort 2 Day 1: APX001 1000 mg IV BID over a 3-hour infusion; Day 24: APX001 1000 mg IV BID over a 3-hour infusion.
  Other Names: Fosmanogepix
Drug: Itraconazole — Cohort 1 Days 15-30: itraconazole 200 mg oral solution QD.
  Other Names: Sporanox
  Arms: Cohort 1
Drug: Rifampin — Cohort 2 Days 15-33: rifampin 600 mg oral QD.
  Other Names: Rifampicin
  Arms: Cohort 2

SUMMARY:
This is a Phase 1, open-label study to evaluate the drug-drug interaction potential of a strong CYP3A4 inhibitor (itraconazole) and a pan-CYP inducer (rifampin) on APX001 in two parallel groups of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal or surgically sterile, or
* Women of childbearing potential must agree to avoid pregnancy during the study and to use contraception, or abstinence, at least 2 weeks before the start of study drug administration until 3 months after the last dose of study drug.
* Male subjects must agree to use barrier contraception, or commit to abstinence, from first Admission to the clinic until 3 months after the last dose of study drug.
* Body mass index (BMI): 18.0 to 32.0 kg/m sq, inclusive
* Weight: >= 50 kg
* Screening hematology, clinical chemistry, coagulation, and urinalysis consistent with overall good health
* Able to understand and comply with the requirements of the study, willing to return for all clinic visits, including confinement periods, and complete all study-related procedures Willing and able to provide written informed consent.

Exclusion Criteria:

* Having any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, ,gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential.
* History or presence of malignancy within the past year. Subjects who have been successfully treated with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled.
* Active acute or chronic infection, including, but not limited to: upper airway infection, urinary tract infection, or skin infection within 30 days preceding entry into the study.
* Significant and/or acute illness within 5 days prior to the first study drug administration that may impact safety assessments, in the opinion of the Investigator.
* Participation in an investigational drug study within 60 days prior to the first study drug administration in the current study. Participation in more than 3 other drug studies in the 10 months prior to the first study drug administration in the current study.
* Use of any prescription medication within 14 days prior to the planned first study drug administration and throughout the study (excluding female contraception).
* Use of any non-prescription or over-the-counter medications within 7 days prior to the planned first study drug administration and throughout the study. This includes all vitamins, other herbal supplements, or remedies.
* Taking any drug or herbal CYP3A modulator (e.g. erythromycin; St. John's Wort) within 4 weeks (or 5 half-lives, whichever is longer) or any other nutrients known to modulate CYP3A activity (e.g. grapefruit juice; Seville orange) within 2 weeks prior to the first Admission.
* History of tobacco or any nicotine-containing product or device use within the past 3 months prior to the planned first study drug administration
* History of alcohol or substance abuse based on Investigator's judgment, within the past 12 months prior to the planned first study drug administration
* Concurrent social conditions (e.g. drugs-of-abuse, alcohol use of more than 24 units per week) that may potentially interfere with the subject's compliance with the protocol
* History of clinically significant allergic drug reactions
* Clinically significant physical examination, vital signs, laboratory safety test, or electrocardiogram (ECG) abnormalities
* Donation or loss of more than 100 mL of blood within 60 days prior to the first study drug administration. Donation or loss of more than 1.5 liters of blood (for male subjects) or more than 1.0 liter of blood (for female subjects) in the 10 months prior to the first study drug administration in the current study.
* Positive results on any of the following screening laboratory tests: serum pregnancy test, urine alcohol test, urine drugs-of-abuse (including cotinine), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
* Prior exposure to APX001
* Known allergy to corn or corn products or any inactive components of the study drug
* Known hypersensitivity to culprit drugs (itraconazole or rifampin).

Additional Exclusion Criteria for Cohort 2:

* Diagnosis or suspected of having porphyria or having first-degree relatives diagnosed or suspected of having porphyria.
* Unwilling not to use contact lenses for the duration of rifampin dosing (Day 15 to Day 33 for Cohort 2) until 7 days after the last dose of rifampin (subjects in Cohort 2 may resume wearing contact lenses on Day 40).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of APX001/APX001A as measured by area under the plasma concentration-time curve (AUC) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by maximum observed plasma concentration (Cmax) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by time to attain maximum observed plasma concentration (Tmax) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by terminal elimination rate constant (λz) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by terminal elimination half-life (t1/2) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by total clearance (CL) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks
Pharmacokinetics of APX001/APX001A as measured by the volume of distribution during the terminal phase (Vz) after multiple doses of a CYP3A4 inhibitor, itraconazole (oral solution) or multiple doses of a pan-CYP inducer, oral rifampin. | 6 weeks

SECONDARY OUTCOMES:
Number of subjects experiencing and frequency of occurrence of adverse events as rated by CTCAE v5.0 after dosing with APX001 IV alone and when co-administered with itraconazole (oral solution) or oral rifampin. | 6 weeks
Occurrence and magnitude of clinical lab test values outside the normal range, clinically significant, and differing from baseline results after dosing with APX001 IV alone and when co-administered with itraconazole (oral solution) or oral rifampin. | 6 weeks
  The following parameters will be measured:
  * Clinical chemistry (serum quantitatively): total bilirubin, direct (conjugated) bilirubin, indirect (unconjugated) bilirubin (calculated), alkaline phosphatase, gamma-GT, ASAT, ALAT, LDH, p-amylase, lipase, CPK, creatinine, eGRF, urea, uric acid, cholesterol, triglycerides, total protein, albumin, globulin, glucose, inorganic phosphate, sodium, potassium, calcium, chloride, and bicarbonate.
  * Hematology (blood quantitatively): leukocytes, erythrocytes, hemoglobin, hematocrit, thrombocytes, partial automated absolute differentiation: lymphocytes, monocytes, eosinophils, basophils, neutrophils, MCV, MCH, and MCHC.
  * Coagulation (blood quantitatively): PT, aPTT, and fibrinogen.
  * Urinalysis (urine qualitatively): color, protein, glucose, bilirubin, urobilinogen, ketones, blood, pH, specific gravity, and leukocytes.
Occurrence of abnormal vital signs after dosing with APX001 IV alone and when co-administered with itraconazole (oral solution) or oral rifampin. | 6 weeks
  Systolic and diastolic blood pressure and pulse will be recorded after the subject has been resting supine or semi-recumbent for at least 5 minutes. Body temperature and respiratory rate will be measured subsequently.
Occurrence of abnormal, clinically significant results from 12-lead ECGs after dosing with APX001 IV alone and when co-administered with itraconazole (oral solution) or oral rifampin. | 6 weeks
  The following ECG parameters will be recorded: heart rate, PR interval, QRS duration, QT interval, and QTc interval (Fridericia's).
Occurrence of changes in physical examinations which differ from baseline after dosing with APX001 IV alone and when co-administered with itraconazole (oral solution) or oral rifampin. | 6 weeks
  Physical examination will include: general appearance; skin/subcutaneous tissue; head; ears, nose, throat; neck and thyroid; thorax; lungs; cardiovascular; lymph nodes; abdomen; musculoskeletal; and neurological.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (2):
- Netherlands (2):
  - PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen
  - PRA-EDS, Groningen

REFERENCES:
- [Derived] Hodges MR, van Marle S, Kramer WG, Ople E, Tawadrous M, Jakate A. Phase 1 drug-drug interaction study to assess the effect of CYP3A4 inhibition and pan-CYP induction on the pharmacokinetics and safety of fosmanogepix in healthy participants. Antimicrob Agents Chemother. 2024 Jun 5;68(6):e0165023. doi: 10.1128/aac.01650-23. Epub 2024 May 17. PMID 38757982